CLINICAL TRIAL: NCT04065984
Title: BiCyCLE: Neuro-Muscular Electrical Stimulation (NMES) and Its Effect on Changes in Body Composition Following Surgery for Locally Advanced Rectal Cancer - a Single Centre Double Blind Randomised Controlled Phase II Clinical Trial
Brief Title: Body Composition Manipulation in CoLorectal cancEr (BiCyCLE): Neuromuscular Electrical Stimulation (NMES)
Acronym: BiCyCLE-NMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 242022
Record Dates: First submitted 2019-04-03; First posted 2019-08-22 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Rectal Cancer; Colorectal Cancer; Colon Cancer; Colo-rectal Cancer; Sarcopenia; Sarcopenic Obesity; Advanced Cancer; Recurrent Rectal Cancer
Keywords: Rectal Cancer; Colorectal Cancer; Recurrent Rectal Cancer; Advanced Rectal Cancer; Myopenia; Sarcopenia; Myosteatosis
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will either receive a device providing active treatment levels of stimulation or a placebo device providing sub therapeutic electrical stimulation.
  The main outcome is change in muscle mass of CT at 3 to 6 months. These scans will be assessed by a radiologist using automated software, the radiologist is blinded to which trial arm the patient was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-Muscular electrical stimulation treatment arm (Experimental): Active muscle stimulation with a view that this will lead to muscle preservation through muscle fibre recruitment
  Interventions: Device: Microstim 2v2 Stimulator
- Neuro-Muscular electrical stimulation Placebo arm (Sham Comparator): Stimulator set at a sub therapeutic threshold so as to not recruit muscle fibres
  Interventions: Device: Microstim 2v2 Stimulator

INTERVENTIONS:
Device: Microstim 2v2 Stimulator — Neuro-muscular electrical stimulator portable device (9v battery) connected to the skin participant over the muscle body of choice using self adhesive electro-gel pads. Treatment devices and placebo devices.

SUMMARY:
Muscle is lost as part of the rectal cancer disease process. Surgery to treat rectal cancer and its subsequent immobility leads to increased muscle loss. Neuromuscular electrical stimulation (NMES) has been shown in previous studies in the critically ill to maintain muscle mass. The investigators aim to examine whether NMES use in the pre and postoperative setting preserves muscle mass, speeds up recovery and improves outcomes in advanced rectal cancer patients undergoing curative surgery. This is a phase II double blind randomised controlled clinical trial.

DETAILED DESCRIPTION:
Myopenia (muscle wasting) occurs as part of the disease process of colorectal cancer, when coupled with the physiological demands and immobility of major surgery there is an even more profound loss in muscle mass.

Evidence suggests that patients who have greater muscle mass and better muscle quality have better post operative outcomes, fewer complications and longer survival. Patients who have pelvic surgery (complex major surgery to remove some or all the pelvic organs involved in the local spread cancer) for locally advanced rectal cancer (cancer of the last part of the large bowel) are highly immobile post operatively.

The investigators are planning to stimulate the thigh and back muscles pre and post operatively in patients undergoing surgery for locally advanced rectal cancer using a device known as a neuromuscular electrical stimulator (NMES). This device mimics exercise in patients, who are unable to exercise fully. The investigators hypothesise that this will prevent the muscle loss normally seen in advanced cancer patients and even, potentially, increase muscle bulk. The investigators will compare this patient group to a control group of patients who are having the same surgery but will use a placebo stimulation protocol. The investigators will compare short and long term outcomes, differences in inflammation and quality of life in both these patient groups.

Neuro-Muscular Electrical Stimulation has been used successfully to help provide physiotherapy in critically ill patients, in earlier studies it has shown preservation of muscle in cancer patients too.

The investigators want to identify whether NMES, as an adjunct to standard parenteral nutritional support and physiotherapy, can help maintain or even increase lean body mass and exert the anti-inflammatory effect of exercise. We want to see if using this device improves quality of life post operatively and improves patient outcomes.

The purpose of this study is to see whether muscle bulk can be preserved and muscle quality maintained in partially immobile post operative advanced rectal cancer patients. This will be done by using a neuromuscular electrical stimulator (NMES) device called a Microstim 2v2 (Odstock Medical Ltd, Salisbury, UK). The investigators are doing this because it is known from previous research that patients with more muscle and better quality muscle have better outcomes following colorectal cancer surgery. It is also known from studies in the critically ill that NMES can successfully increase muscle and can act as a surrogate for exercise. The investigators aim to identify whether muscle bulk and quality can be increased and improved in these patients and indeed, whether this reduces inflammation, improves recovery, outcomes and Quality of Life. the investigators also want to see if patients find the device easy and acceptable to use.

This will be run as a single centre double blind randomised controlled phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above
* Male or female
* Primary or recurrent locally advanced rectal cancer amenable to elective radical exenterative surgery
* ASA grade I-III
* Able and willing to consent
* Participation in other concurrent trials is acceptable - following discussion with trial team of both studies.

Exclusion Criteria:

* Lack of patient consent
* Wide spread metastases not amenable to curative resection
* Contraindication to NMES (see appendix 6)
* Pre existing neuromuscular degenerative disease
* Participation in other trials where agreement on participation not made in advance by trial teams
* Patients with solitary colon cancer above the level of the peritoneal reflexion which does not require complex pelvic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean muscle attenuation pre and postoperatively | 2 years
  The difference in mean muscle attenuation (MA) measured in Hounsfield units between the pre- operative and 3 month post-operative CT scan in the NMES treatment group and the placebo NMES group.

SECONDARY OUTCOMES:
CT derived muscle measurements | 6 months
  The difference in Lumbar skeletal Muscle Index (LSMI=height / area of skeletal muscle in cm2 at L3) derived from the third lumbar vertebral axial level of pre and 3 to 6 month postoperative CT scans using SliceOmatic software version 5.0 with ABACS L3 Plug-in automation tool.
CT derived fat measurements | 6 months
  The difference in Visceral Adipose Tissue (cm2) derived from the third lumbar vertebral axial level of pre and 3 to 6 month postoperative CT scans using SliceOmatic software version 5.0 with ABACS L3 Plug-in automation tool.
Pre and Post-operative systemic inflammation | 6 months
  C-reactive protein (CRP)
Pre and Post-operative systemic cellular immune response | 6 months
  Neutrophil to Lymphocyte ratio (NLR)
Short-term post surgical complications | 6 months
  Clavien-Dindo Score for postoperative complications (1-5)
Hospital Stay | 6 months
  Length of hospital stay in days
Quality of Life (General - EQ- 5D- 5L) | 2 years
  EuroQol 5-level EQ-5D version, consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  Five dimensions are analysed: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored from 1 to 5 ranging from: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The patient ticks a box corresponding to indicate their status within each dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  Post-operative quality of life at 6 months and 12 months following surgery using the validated quality of life questionnaire ED-5Q-5L will be assessed as described above.
Quality of Life (Colorectal specific - EORTC QLQ - CR29) | 2 years
  European Organisation for Research and Treatment of Cancer (EORTC) colorectal QoL module QLQ-CR29. The QLQ-CR29 contains 4 multi item scales and 19 single items assessing common symptoms and problems in colorectal cancer. The scales and single item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problems.
  Post-operative quality of life at 6 months and 12 months following surgery using the validated quality of life questionnaire EORTC QLQ - CR29
Function | 6 months
  Function as assessed by the Berg Balance scale, sit-to-stand and 6-minute walk test at baseline and approximately 3 months following surgery
Thigh circumference | 2 years
  Difference in thigh circumference both legs (at 15cm above the superior pole of the patella) preoperatively and at 3 month postoperatively.
Bio-impedance measures of body composition | 2 years
  Bio-impedance analysis (BIA) metrics at set time points (baseline, day two post operatively, day twenty-eight post operatively (if in hospital) day of discharge, first post-operative follow u appointment.
Device satisfaction | 10 weeks
  Patient satisfaction with using the NMES device.
Device dose response | 2 years
  Dose response to NMES utilising the patient compliance diary and CT derived data.
Sequential CT changes in body composition | 5 years
  Sequential changes measure on CT over a 5-year follow-up period following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Pring, BSc MRCS, Principal Investigator — LNWUH NHS Trust
Locations (1):
- London North West University Healthcare NHS Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan at present for data sharing however patients will consent for fully anonymised data sharing to occur. No identifiable information will be shared.

REFERENCES:
- [Background] Malietzis G, Currie AC, Johns N, Fearon KC, Darzi A, Kennedy RH, Athanasiou T, Jenkins JT. Skeletal Muscle Changes After Elective Colorectal Cancer Resection: A Longitudinal Study. Ann Surg Oncol. 2016 Aug;23(8):2539-47. doi: 10.1245/s10434-016-5188-1. Epub 2016 Mar 22. PMID 27006127
- [Background] Malietzis G, Johns N, Al-Hassi HO, Knight SC, Kennedy RH, Fearon KC, Aziz O, Jenkins JT. Low Muscularity and Myosteatosis Is Related to the Host Systemic Inflammatory Response in Patients Undergoing Surgery for Colorectal Cancer. Ann Surg. 2016 Feb;263(2):320-5. doi: 10.1097/SLA.0000000000001113. PMID 25643288
- [Background] Malietzis G, Currie AC, Athanasiou T, Johns N, Anyamene N, Glynne-Jones R, Kennedy RH, Fearon KC, Jenkins JT. Influence of body composition profile on outcomes following colorectal cancer surgery. Br J Surg. 2016 Apr;103(5):572-80. doi: 10.1002/bjs.10075. PMID 26994716
- [Background] Grande AJ, Silva V, Maddocks M. Exercise for cancer cachexia in adults: Executive summary of a Cochrane Collaboration systematic review. J Cachexia Sarcopenia Muscle. 2015 Sep;6(3):208-11. doi: 10.1002/jcsm.12055. Epub 2015 Jul 7. PMID 26401466
- [Background] Maddocks M, Lewis M, Chauhan A, Manderson C, Hocknell J, Wilcock A. Randomized controlled pilot study of neuromuscular electrical stimulation of the quadriceps in patients with non-small cell lung cancer. J Pain Symptom Manage. 2009 Dec;38(6):950-6. doi: 10.1016/j.jpainsymman.2009.05.011. PMID 19748761
- [Derived] Pring ET, Gould LE, Malietzis G, Lung P, Bharal M, Fadodun T, Bassett P, Naghibi M, Taylor C, Drami I, Chauhan D, Street T, Francis NK, Athanasiou T, Saxton JM, Jenkins JT; BiCyCLE Research Group. BiCyCLE NMES-neuromuscular electrical stimulation in the perioperative treatment of sarcopenia and myosteatosis in advanced rectal cancer patients: design and methodology of a phase II randomised controlled trial. Trials. 2021 Sep 15;22(1):621. doi: 10.1186/s13063-021-05573-2. PMID 34526100